CLINICAL TRIAL: NCT05801835
Title: A Randomized, Open-label, Two-period, Two-way Crossover Bioequivalence Study of Two (Cytarabine: Daunorubicin) Liposome for Injection in Elderly AML Subjects
Brief Title: A Bioequivalence Study of (Cytarabine: Daunorubicin) Liposome for Injection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: CSPC Zhongnuo Pharmaceutical (Shijiazhuang) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HC1702-003
Record Dates: First submitted 2023-03-13; First posted 2023-04-06 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Liposomes; Injections; CPX-351

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence A (T-R) (Experimental): (cytarabine: daunorubicin) liposome for injection followed by Vyxeos
  Interventions: Drug: (cytarabine: daunorubicin) liposome for injection; Drug: Vyxeos
- Sequence B (R-T) (Experimental): Vyxeos followed by (cytarabine: daunorubicin) liposome for injection
  Interventions: Drug: Vyxeos; Drug: (cytarabine: daunorubicin) liposome for injection

INTERVENTIONS:
Drug: (cytarabine: daunorubicin) liposome for injection — Be given intravenously at 65U/m^2 on days 1 and day3 of the first cycle of induction.
  Arms: Sequence A (T-R)
Drug: Vyxeos — Be given intravenously at 65U/m^2 on days 1 and day3 of the first cycle of induction.
  Other Names: CPX-351
  Arms: Sequence B (R-T)
Drug: (cytarabine: daunorubicin) liposome for injection — Be given intravenously at 65U/m^2 on days 1 and day3 of the second cycle of induction.
  Arms: Sequence B (R-T)
Drug: Vyxeos — Be given intravenously at 65U/m^2 on days 1 and day3 of the second cycle of induction.
  Other Names: CPX-351
  Arms: Sequence A (T-R)

SUMMARY:
The purpose of this study is to determine the bioequivalence of (cytarabine: daunorubicin) liposome for injection and Vyxeos in elderly acute myeloid leukemia (AML) subjects.

DETAILED DESCRIPTION:
This is a multi-center, randomized, open-label, two-period, two-sequence, two-way crossover bioequivalence study of (cytarabine: daunorubicin) liposome for injection manufactured by CSPC Zhongnuo Pharmaceutical Technology Co., Ltd compared with Vyxeos manufactured by Jazz Pharmaceuticals, Inc. in elderly AML subjects. Patients who have achieved CR/CRi after induction treatment will be randomized to sequence A (T-R): (cytarabine: daunorubicin) liposome on C1D1 and C1D3/ Vyxeos on C2D1 and C2D3 or sequence B(R-T): Vyxeos on C1D1 and C1D3/ (cytarabine: daunorubicin) liposome on C2D1 and C2D3. Randomization will be in a 1:1 ratio. Forty to sixty subjects will be enrolled to ensure 36 evaluable subjects.

Serial blood samples for determination of liposomal encapsulated cytarabine and liposomal encapsulated daunorubicin plasma concentration for PK analysis will be obtained in each cycle.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand the study and voluntarily sign informed consent.
2. Male or female between 55-75 years of age (inclusive).
3. Subjects diagnosed with acute myeloid leukemia according to "The 2016 revision to the World Health Organization classification of myeloid neoplasms and acute leukemia" who haven't been treated or who have achieved complete remission (CR) or complete remission with incomplete blood count recovery (CRi) after preceding induction therapy.
4. Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
5. Adequate hematopoietic, renal and liver function.
6. Cardiac function (LVEF) ≥ 50% and QTcF (Fridericia's) for male<450 ms, for female<470 ms at screening.
7. Women of childbearing potential should agree to use contraceptive measures (such as IUD, contraceptive or condom) during the study and within 6 months after the end of the study.

Exclusion Criteria:

1. Subjects who are diagnosed as acute promyelocytic leukemia.
2. Subjects with clinical evidence of active CNS leukemia.
3. Subjects with any other active malignancy expect for those have been cured (basal cell carcinoma, superficial bladder cancer, cervical cancer in situ, carcinoma in situ of breast or prostate cancer with Gleason score <6).
4. For subjects with induction remission who go directly to randomisation, their antitumour drug elution is required prior to the first dose in the consolidation phase for a minimum of 5 half-lives or 4 weeks, whichever is shorter.
5. Subjects with a history of any major surgery or radiation therapy within 4 weeks prior to the first dose.
6. Subjects with active cardiovascular disease within 6 months prior to the first dose.
7. Subjects with severe hemorrhagic disorders or diseases may cause spontaneous bleeding.
8. Subjects with active or history of cerebrovascular disease, such as stroke, cerebral hemorrhage within 6 months prior to the first dose.
9. Subjects with severe pulmonary disease within 2 weeks prior to the first dose.
10. Subjects with active or uncontrolled infection.
11. Subjects with previous cumulative exposure to anthracyclines >302 mg/m^2 daunorubicin (or equivalent drug equivalent dose level).
12. Subjects with hypersensitivity to liposomal products.
13. Subjects with a history of Wilson's disease or other copper-metabolism disorder.
14. Subjects with known HIV, hepatitis B or hepatitis C infection.
15. Participation in another clinical trial or treatment with any investigational drug within 28 days of study start
16. Female subjects who are pregnant, breast-feeding, or who are likely to become pregnant during the study.
17. Any subject whom the Investigator believes will not be a good candidate for the study.

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-08-25 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Maximum (peak) plasma drug concentration (Cmax) of daunorubicin cytarabine liposomes | 30 minutes before administration and 1.5, 2, 5,9,24,48,72,120,168hours after administration of Day 1.
  Maximum (peak) plasma drug concentration is a Pharmacokinetic parameter
Area under the plasma concentration versus time curve calculated from 0 to 48h post administration (AUC0-48h) of daunorubicin cytarabine liposomes | 30 minutes before administration and 1.5, 2, 5,9,24,48,72,120,168hours after administration of Day 1
  Area under the plasma concentration-time curve from time zero to time 48 hours is a Pharmacokinetic parameter

SECONDARY OUTCOMES:
Maximum (peak) plasma drug concentration (Cmax) of free daunorubicin and cytarabine | 30 minutes before administration and 1.5, 2, 5,9,24,48,72,120,168hours after administration of Day 1.
  Maximum (peak) plasma drug concentration is a Pharmacokinetic parameter
Area under the plasma concentration versus time curve calculated from 0 to 48h post administration (AUC0-48h) of free daunorubicin and cytarabine | 30 minutes before administration and 1.5, 2, 5,9,24,48,72,120,168hours after administration of Day 1.
  Area under the plasma concentration-time curve from time zero to time 48 hours is a Pharmacokinetic parameterencapsulated and toal cytarabine and daunorubicin after Day 3 treatment of each period.
Maximum (peak) plasma drug concentration (Cmax) of total daunorubicin and cytarabine | 30 minutes before administration and 1.5, 2, 5,9,24,48,72,120,168hours after administration of Day 1.
  Maximum (peak) plasma drug concentration is a Pharmacokinetic parameter
Area under the plasma concentration versus time curve calculated from 0 to 48h post administration (AUC0-48h) of total daunorubicin and cytarabine | 30 minutes before administration and 1.5, 2, 5,9,24,48,72,120,168hours after administration of Day 1.
  Area under the plasma concentration-time curve from time zero to time 48 hours is a Pharmacokinetic parameterencapsulated and toal cytarabine and daunorubicin after Day 3 treatment of each period.
Incidence of treatment-emergent adverse events (TEAEs) | Up to 35 calendar days after the last administration of the investigational product.
Complete remission rate | Up to 1 year.
  Proportion of subjects with complete remission
Composite remission rate | Up to 1 year.
  Proportion of subjects with complete response (CR) or complete response with incomplete count recovery (CRi)
Relapse-free survival | Up to 3 years.
  From the date of remission to the date of relapse after CR/CRi, or death, whichever occurs first.
Proportion of subjects who achieve complete remission with MRD negativity | Up to 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Jianxiang Wang, MD, Principal Investigator — Chinese Academy of Medical Sciences & Peking Union Medical College
Locations (1):
- Institute of Hematology and Hospital of Blood Disease, Chinese Academy of Medical Sciences, Tianjin, China